CLINICAL TRIAL: NCT01174823
Title: Safety and Efficacy of Bepotastine Besilate Ophthalmic Solution in Seasonal Allergic Conjunctivitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S00041
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bepotastine Besilate Ophthalmic Solution (Experimental)
  Interventions: Drug: bepotastine besilate ophthalmic solution
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo comparator ophthalmic solution

INTERVENTIONS:
Drug: bepotastine besilate ophthalmic solution — sterile ophthalmic solution
  Arms: Bepotastine Besilate Ophthalmic Solution
Drug: placebo comparator ophthalmic solution — sterile ophthalmic solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to study the safety and efficacy of bepotastine besilate ophthalmic solution in allergic conjunctivitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 12 years of age and older with 2-year history of allergic conjunctivitis

Exclusion Criteria:

* No active ocular or nasal infection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

REFERENCES:
- [Derived] Carr WW, Nayak AS, Ratner PH, Gow JA, McNamara TR, Williams JI; Bepotastine Besilate Ophthalmic Solution 1.5% (Bepreve) Study Group. Efficacy of bepotastine besilate ophthalmic solution 1.5% for seasonal allergic conjunctivitis: a randomized, placebo-controlled, natural exposure, clinical trial. Allergy Asthma Proc. 2013 May-Jun;34(3):247-54. doi: 10.2500/aap.2013.34.3671. PMID 23484763

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo comparator ophthalmic solution: sterile ophthalmic solution administered twice a day
- Bepotastine Besilate Ophthalmic Solution: bepotastine besilate ophthalmic solution: sterile ophthalmic solution administered twice a day
Period: Overall Study
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Started | 122 | 123
Completed | 115 | 119
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (15.0) | 38.7 (13.8) | 40.1 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 71 | 153
  Male | 40 | 52 | 92

OUTCOME MEASURES:

1. Primary Outcome: Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) - Mean Change in Total Score
Description: Responses to questions relating to symptoms and daily activities in the RQLQ were provided for 28 questions encompassing the 7 major domains of activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional state. Each response to an RQLQ question was provided on a scale of 0-6 units, where 0 = not troubled/none of the time and 6 = extremely troubled/all of the time. The minimum total score was 0 units and the maximum total score was 42 units, with higher score indicating decreased quality of life due to rhinoconjunctivitis.
Time Frame: Baseline, 14 days
Population: The per protocol population included randomized participants with no major protocol violations, who had at least 80% dosing compliance during the 2-week dosing period and at least 85% compliance in providing nasal and ocular symptom grades in the Subject Diary, and who completed the RQLQ at Day 0 and Day 14 (+2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
score on a scale | -1.18 (1.24) | -1.17 (1.27)

2. Secondary Outcome: Mean Change From Baseline for Twice Daily (BID) Averaged Reflective Ocular Itching Scores Over the Treatment Period
Description: Ocular itching was graded on a 4-point scale (0-3 units; 0=Absent, 1=Mild, 2=Moderate, 3=Severe) twice daily in the Screening Diary (Day -7 to Day -1) and the Subject Diary (Day 0 prior to first dose through Day 13).
Time Frame: Baseline, 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
score on a scale | -0.54 (0.58) | -0.71 (0.65)

3. Secondary Outcome: Mean Change From Baseline for Twice Daily (BID) Averaged Instantaneous Ocular Redness Scores Over the Treatment Period
Description: Ocular redness each was graded on a 4-point scale (0-3 units; 0=Absent, 1=Mild, 2=Moderate, 3=Severe) twice daily in the Screening Diary (Day -7 to Day -1) and the Subject Diary (Day 0 prior to first dose through Day 13).
Time Frame: Baseline, 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
score on a scale | -0.45 (0.61) | -0.62 (0.57)

4. Secondary Outcome: Mean Change From Baseline for Twice Daily (BID) Averaged Proportion of Tearing Episodes Over the Treatment Period
Description: Individual nasal symptoms and ocular itching and redness each were graded on a 4-point scale (0-3 units; 0=Absent, 1=Mild, 2=Moderate, 3=Severe) BID in the Screening Diary (Day -7 to Day -1) and BID in the Subject Diary (Day 0 prior to first dose through Day 13). Tearing was scored from Day 0 as either absent or present at the same time as nasal and other ocular symptoms were graded. The proportion of participants was calculated and then then average of the proportions.
Time Frame: Baseline, 14 days
Population: The per protocol population included randomized participants with no major protocol violations, who had at least 80% dosing compliance during the 2-week dosing period, who had at least 85% compliance in providing nasal and ocular symptom grades in the Subject Diary, and who completed the questionnaire at Day 0 and Day 14 (+2).
Measure: Mean (Standard Deviation); unit: tearing episodes
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
tearing episodes | -0.15 (0.244) | -0.18 (0.269)

5. Secondary Outcome: Mean Change From Baseline for Twice Daily (BID) Averaged Reflective Total Nasal Symptom Scores Over the Treatment Period
Description: Individual nasal symptoms of rhinorrhea, nasal congestion, nasal itching, and sneezing each were each graded on a 4-point scale (0-3 units; 0=Absent, 1=Mild, 2=Moderate, 3=Severe) twice daily in the Screening Diary (Day -7 to Day -1) and the Subject Diary (Day 0 prior to first dose through Day 13). The minimum Total Nasal Symptom Score (TNSS) was 0 units and the maximum TNSS corresponding to multiple individual nasal symptoms scored as severe was 12 units
Time Frame: Baseline, 14 days
Population: The per protocol population included randomized participants with no major protocol violations, who had at least 80% dosing compliance during the 2-week dosing period and at least 85% compliance in providing nasal and ocular symptom grades in the Subject Diary, and who completed the questionnaire at Day 0 and Day 14 (+2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
score on a scale | -1.73 (1.94) | -2.08 (2.06)

6. Secondary Outcome: Global Therapeutic Response Rating - Participant Assessed
Description: Participants were asked if they felt that they had experienced improvement in allergy symptoms after therapy. Participant assessed global therapeutic response rating: categories that the participant could select were 'no change', 'slight improvement', 'improved', or 'marked improvement'.
Time Frame: 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
Participants
  Improved or Marked Improvement | 24 | 27
  Any Improvement | 64 | 72

7. Secondary Outcome: Global Therapeutic Response Rating - Investigator Assessed
Description: Investigators were asked if they felt that the participant had experienced improvement in allergy symptoms after therapy. Investigator assessed global therapeutic response rating: categories that the investigator could select were 'no change', 'slight improvement', 'improved', or 'marked improvement'.
Time Frame: 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
Number analyzed (Participants) | 107 | 109
Participants
  Improved or Marked Improvement | 16 | 29
  Any Improvement | 56 | 70

ADVERSE EVENTS:
Time Frame: 14 days
Description: The analysis population for the adverse events was randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | Bepotastine Besilate Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/123
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/123
Other Adverse Events (participants affected / at risk) | 1/121 | 10/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Bepotastine Besilate Ophthalmic Solution (N=123)
Localized infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Bepotastine Besilate Ophthalmic Solution (N=123)
Mild taste following instillation (General disorders) | 1 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.